CLINICAL TRIAL: NCT00444639
Title: Phase II Multi-Centric, Randomised, Open-label, Parallel-Group Study to Assess the Non-inferiority of Pamorelin® 11,25mg SC Injected Versus Pamorelin® 11,25mg IM Injected in Patients Suffering From Advanced Prostate Cancer
Brief Title: Study to Assess the Non-inferiority of Pamorelin® 11,25mg SC Injected Versus Pamorelin® 11,25mg IM Injected in Patients Suffering From Advanced Prostate Cancer (PAMOJECT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-48-52014-142; 2005-005058-31 (EudraCT Number)
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

ARMS (2):
- 1 (Experimental): triptorelin 11.25mg given 12 weekly by subcutaneous formulation
  Interventions: Drug: Triptorelin (Decapeptyl®)
- 2 (Active Comparator): triptorelin 11.25mg given 12 weekly by intramuscular injection
  Interventions: Drug: Triptorelin (Decapeptyl®)

INTERVENTIONS:
Drug: Triptorelin (Decapeptyl®) — Two injections of 11.25mg given every 12 weeks

SUMMARY:
The active ingredient of Pamorelin® 11,25 mg is Triptorelin. Triptorelin is a substitute for a natural hormone produced in the body called Gonadotrophin-releasing hormone (GnRH). GnRH is a hormone secreted by hypothalamus (a gland located in brain) and controls the production of sex hormones (eg testosterone in men) in other organs in the body. The growth of prostate cancer cells, one of the most common cancers in men, is induced by the hormone testosterone. Hormonotherapy is one of treatments available to treat this type of disease by controlling the testosterone serum level. Pamorelin® 11,25 mg is normally injected in the muscle but this type of injection is not suitable for every patient. Therefore the primary purpose of this study is to assess the non-inferiority of the 12-week triptorelin formulation Pamorelin® 11,25 mg administered via subcutaneous (SC) injection as compared to Pamorelin® 11,25 mg administered via standard intramuscular (IM) injection based on the percentage of patients presenting a testosterone level ≤ 50 ng/dl at week 24.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven prostate cancer, locally advanced or metastatic and scheduled to receive hormonal deprivation therapy
* Life expectancy of more than 9 months
* Documented testosterone levels of ≥ 125 ng/dl measured by any laboratory or on site within the previous 6 months

Exclusion Criteria:

* Has a history of hypersensitivity to the Investigational Medicinal Product or drugs with a similar chemical structure
* Has previously received a GnRH analogue, estrogens or a steroidal anti -androgen within the last year preceding the study
* Concomitant anti-coagulation treatment
* Patient who underwent an orchidectomy or who is scheduled to receive an orchidectomy during the course of this study
* Patient with known spinal medullar compression

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving a plasma testosterone level ≤ 50 ng/dl (1,7 nmol/l). | Week 24

SECONDARY OUTCOMES:
Patient acceptability of the injection; the pain experienced during injection, scored by means of a Visual Analogue Scale (VAS). | Measured at baseline and 12 weeks
Care giver acceptability of the administration of the injection by means of a Visual Analogue Scale (VAS). | Measured at baseline and 12 weeks
Percentage of patients achieving a plasma testosterone level ≤ 50 ng/dl (1,7 nmol/l). | Measured at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (15):
- Netherlands (15):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - AMC Amsterdam, Amsterdam
  - Alysis Zorggroep Loc. Rijnstate, Arnhem
  - Maasziekenhuis Pantein, Boxmeer
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - St. Anna Ziekenhuis Geldrop, Geldrop
  - Groen Hart Ziekenhuis, Gouda
  - Ziekenhuis Hilversum, Hilversum
  - Westfries Gasthuis Hoorn, Hoorn
  - Diaconessenhuis Leiden, Leiden
  - Erasmus MC Rotterdam, Rotterdam
  - Antonius Ziekenhuis, Sneek
  - UMC Utrecht, Utrecht
  - Albert Schweitzer Ziekenhuis, Zwijndrecht